CLINICAL TRIAL: NCT04966286
Title: The Effectiveness of Applying Multimedia on Self-Care and Quality of Life in Patient With Enterostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7425
Record Dates: First submitted 2021-06-28; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Multimedia Learning Education; Self-care; Quality of Life; Enterostomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional education service program (Placebo Comparator): received only standard enterostomy care brochure
  Interventions: Other: multimedia education
- multimedia education service program (Experimental): received multimedia education service program introduction
  Interventions: Other: multimedia education

INTERVENTIONS:
Other: multimedia education — The MLEP intervention was based on a literature review of prior research on the content and format of self care related multimedia education programmes

SUMMARY:
This report was an effective evaluation of using multimedia educational program for self-care and quality of life in patients with a stoma at postoperative and established a simple threshold for enterostomy self-care skills.

DETAILED DESCRIPTION:
In a systematic review, evaluated the effectiveness of multimedia education program (MLEP) and confirmed that MLEP reduced cost significantly and improved patient participation in enterostomy care and self-care ability. However, research was insufficient for whether a multimedia education program (MLEP) interventions can improve patient self-care and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 20
* Operation with ostomy

Exclusion Criteria:

* Dementia, mental illness, and central nervous system diseases
* Unable self-care
* Visual or hearing impairs

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
self-care ability | One and a half years
  Assessment scale of self-care ability of enterostomy care was a quantitative scale for nursing staff to evaluate self-care skills in patients with enterostomy. It consisted of 7 items related to: Prepare items, removing the pouching system, measuring the enterostomy diameter, adjusting the size of the enterostomy diameter in a new stoma appliance, skin care, fitting a new enterostomy appliance, and emptying procedure. Each skill was rated on a 4-point scale: Likert scale (1: not at all, 2: some, 3: quite a lot, 4: very much).
  Higher scores indicated that patient had a higher level of self-care skills for changing enterostomy pouching system

SECONDARY OUTCOMES:
Promote quality of life | One and a half years
  The Enterostomy quality of life was comprised of 30 questionnaires, it covered seven domains: relations with family and friends, Sleep, activity, sexual activity, social relationship, physiology and psychology. The responses rated on a4-point scale Likert scale (1: extremely, 2: quite a lot, 3: somewhat, 4: not at all). The possible scores range was from 37 to 148. Higher scores indicated that patient had a higher level of quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Hsing Fang Ko, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No